CLINICAL TRIAL: NCT03937206
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Ranging Study to Evaluate the Pharmacokinetics, Safety and Effects of NutriterraTM in Healthy Adult Subjects
Brief Title: Evaluation of the Pharmacokinetics, Safety and Effects of NutriterraTM in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nuseed Americas Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NUSERPD-160001-RPD01
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Healthy
MeSH Terms: interventions — Rapeseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose (Experimental): Low Dose (300mg TG Omega-3) - 1 capsule containing 1000mg NutriterraTM per capsule + 3 capsules containing 1000mg corn oil per capsule
  Interventions: Dietary Supplement: NutriterraTM; Dietary Supplement: Placebo
- Mid Dose (Experimental): Mid Dose (600mg TG Omega-3) - 2 capsules containing 1000mg NutriterraTM per capsule + 2 capsules containing 1000mg corn oil per capsule
  Interventions: Dietary Supplement: NutriterraTM; Dietary Supplement: Placebo
- High Dose (Experimental): High Dose (1200mg TG Omega-3) - 4 capsules containing 1000mg NutriterraTM per capsule
  Interventions: Dietary Supplement: NutriterraTM
- Placebo (Placebo Comparator): Placebo (0mg TG Omega-3) - 4 capsules containing 1000mg corn oil per capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NutriterraTM — Nutriterra 1000mg
  Other Names: Canola Oil
  Arms: High Dose; Low Dose; Mid Dose
Dietary Supplement: Placebo — Corn Oil 1000mg
  Arms: Low Dose; Mid Dose; Placebo

SUMMARY:
The blood lipid profile plays a role in health and disease states and is affected by many genetic and lifestyle factors. On the more extreme side, hyperlipidemia (a condition characterized by hypertriglyceridemia, hypercholesteremia, or both) is a risk factor for coronary heart disease (CHD) 1. CHD is the most common form of cardiovascular disease (CVD); it is characterized by arterial obstructions or blockages, and is a leading cause of heart attacks and strokes 2. Specifically, blood lipids including triglycerides (TG), total cholesterol (TC), low density lipoprotein-cholesterol (LDL-C), and the ratio of TC: high density lipoprotein (HDL) cholesterol, are key modifiable risk factors for CHD. Hyperlipidemia is thought to be caused or promoted by sedentary lifestyle, obesity, or uncontrolled type 2 diabetes 2. Therefore, lifestyle factors, like the modification of dietary lipids to maintain a healthy blood lipid profile are warranted.

There are many beneficial effects of omega-3 fatty acids in terms of cardiovascular disease and the nervous system in general, as well as emerging research on DHA supplementation in acute brain and spinal cord injury. Demand for dietary omega-3's, either through increased fish consumption or through DHA supplementation, is expected to increase, particularly as the baby boomer population adds to the ranks of senior citizens concerned about and/or susceptible to health issues such as dementia and Alzheimer's Disease. Availability of EPA and DHA in circulation is an important parameter in understanding biologic properties of fatty acids.

The purpose of this study is to evaluate the pharmacokinetic characteristics of ascending doses of NutriterraTM, as measured by plasma levels of total EPA, DHA, DPA and ALA under fed conditions. In addition, after a two-week (minimum) washout period, subjects will take product for 16 weeks to evaluate effects on cardiovascular markers as a measure of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years to 80 years (inclusive) at time of screening with suitable veins for cannulation or repeated venipuncture.
* BMI ≥ 18.5 to ≤ 34.9 kg/m2 at the time of Screening
* Female participants of childbearing potential (i.e. not surgically sterilized or post-menopausal greater than one year) must have negative urine pregnancy test and must be using an effective birth control method, defined as:

  * Continuous use of oral or long acting injected contraceptive for at least 2 months prior to study entry, or
  * Use of an intra-uterine device or implantable contraceptive, or
  * Use of double barrier methods of birth control, or
  * Abstinence from heterosexual intercourse
* Willing to avoid alcohol consumption for 24 h prior to every clinic visit
* Willing to avoid moderate to intense exercise 24 h prior to every clinic visit
* Consume less than 200 mg omega-3 per day based on validated Questionnaire
* Agrees to stop taking any vitamins, minerals, or any fatty acid containing dietary/herbal supplements that could potentially interfere with the study endpoints and will be washed out for two weeks prior to study product administration and throughout the study.
* Willing to maintain a stable diet and level of activity throughout the trial.
* Willing to keep a daily journal describing impact of dosage and tolerability.
* Able to comply with all protocol activities.
* Willing and able to provide informed written consent.

Exclusion Criteria:

* Consumption of fish within two weeks prior to the first investigational product administration and for the duration of the study.
* Used canola oil, fish oil, other omega-3 fatty acids (EPA and/or DHA) containing supplements within one (1) month of baseline (Visit 2) or any time during the study, other than the product being evaluated in this study.
* Have a known sensitivity or allergy to canola or any other ingredients in the test products.
* Individuals taking prescription or non-prescription health products that may affect the study endpoint (e.g. corticosteroids, prescription anti-inflammatory drugs, blood lipid-lowering drugs (e.g. statins, fibrates, bile acid exchanger resin, phytosterols, niacin or its analogues, carnitine, etc.) in the previous 6 months.
* Individuals taking any supplements with phytosterols, polyglucosamines (Chitosan) or other lipid-binding ingredients in the previous 3 months.
* Unstable use (i.e. initiation or change in dose) of antihypertensive medications or thyroid hormone replacement medications within 3 months prior to visit 1.
* Use of any weight-loss programs or weight-loss medications (prescription or over-the counter) including, but not limited to, lipase inhibitors, within 6 months prior to visit 1 and throughout the study.
* Pregnancy or lactation, or participant unwilling to take appropriate contraceptives for the duration of the study.
* History of blood clotting disorders or use of coagulation-inhibiting drugs (e.g. warfarin).
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e. Crohn's disease, short bowel, acute or chronic pancreatitis or pancreatic insufficiency).
* Presence of major diseases such as diabetes, endocrine, cardiovascular, renal, or liver disease.
* History of neurological disease (e.g. Parkinson's disease, stroke, traumatic brain injury, etc.).
* History of cancer (excluding non-melanoma skin cancer and basal cell carcinoma) in the past 5 years.
* Uncontrolled hypertension defined as a seated resting systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg.
* Active psychiatric disease (hospitalized within the past 12 months of Screening).
* Documented medical history of immune disorder (such as HIV/aids, hepatitis B or hepatitis C) or positive laboratory results within 28 days of dosing.
* History of a surgical procedure for the treatment of obesity (i.e., gastric bypass, gastric banding).
* Taking potent CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, posaconazole, voriconazole, erythromycin, clarithromycin, telithromycin and nefazodone) within two weeks prior to first investigational product administration and throughout the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
EPA Area Under the Curve | 72 hours
  To determine the pharmacokinetics over a 72-hour period of NutriterraTM at three doses under fed conditions in healthy subjects
DHA Area Under the Curve | 72 hours
  To determine the pharmacokinetics over a 72-hour period of NutriterraTM at three doses under fed conditions in healthy subjects
Triglycerides | 16 weeks
  To evaluate the dose response and effect of NutriterraTM on triglyceride (TG) levels in healthy subjects

SECONDARY OUTCOMES:
Total Cholesterol | 16 weeks
  To determine the effect of daily use of NutriterraTM on total cholesterol
HDL-C | 16 weeks
  To determine the effect of daily use of NutriterraTM on HDL-C
LDL-C | 16 weeks
  To determine the effect of daily use of NutriterraTM on LDL-C
LDL-C/HDL-C ratio | 16 weeks
  To determine the effect of daily use of NutriterraTM on LDL-C/HDL-C ratio
non-HDL-C | 16 weeks
  To determine the effect of daily use of NutriterraTM on non-HDL-C
Omega-3 fatty acid profile in whole blood | 4 weeks
  To determine the effect of daily use of NutriterraTM on whole blood omega-3 fatty acid profile
Omega-3 fatty acid profile in red blood cells | 16 weeks
  To determine the effect of daily use of NutriterraTM on red blood cell omega-3 fatty acid profile
C-reactive protein | 4 and 16 weeks
  To determine the effect of daily use of NutriterraTM on high sensitivity C-reactive protein (hs-CRP)

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrasource, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No